CLINICAL TRIAL: NCT04492020
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Efficacy, Safety, and Tolerability of Oral Ubrogepant in the Acute Treatment of Migraine When Administered During the Prodrome
Brief Title: Study to Evaluate Oral Ubrogepant in the Acute Treatment of Migraine During the Prodrome in Adult Participants
Acronym: UBR Prodrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3110-304-002
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Sequence A (Experimental): Participants randomized to Treatment Sequence A will receive placebo to treat their first qualifying prodrome event and ubrogepant 100 mg to treat their second qualifying prodrome event
  Interventions: Drug: Ubrogepant 100 mg; Drug: Placebo
- Treatment Sequence B (Experimental): Participants randomized to Treatment Sequence B will receive ubrogepant 100 mg to treat their first qualifying prodrome event and placebo to treat their second qualifying prodrome event
  Interventions: Drug: Ubrogepant 100 mg; Drug: Placebo

INTERVENTIONS:
Drug: Ubrogepant 100 mg — For each qualifying prodrome event, 2 compressed tablets containing 50 mg of ubrogepant will be taken orally when the participant is confident that a headache will follow within 1-6 hours
Drug: Placebo — For each qualifying prodrome event, 2 compressed tablets containing placebo will be taken orally when the participant is confident that a headache will follow within 1-6 hours

SUMMARY:
Study to Evaluate the Efficacy, Safety, and Tolerability of Oral Ubrogepant in the Acute Treatment of Migraine When Administered During the Prodrome

ELIGIBILITY:
Inclusion Criteria:

* At least a 1-year history of migraine with or without aura consistent with a diagnosis according to the ICHD-3 (International Classification of Headache Disorders 3rd edition)
* Migraine onset before age 50 years
* By history, the participant's migraines typically last between 4 and 72 hours if untreated or treated unsuccessfully and migraine episodes are separated by at least 48 hours of headache pain freedom
* History of 2 to 8 migraine attacks per month with moderate to severe headache in each of the 3 months prior to the Screening Visit

Exclusion Criteria:

* Difficulty distinguishing migraine headache from tension-type or other headaches
* Participants who overuse medication for migraine defined as use of opioids or barbiturates > 2 days/month, triptans or ergots ≥ 10 days/month, or simple analgesics (eg, aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), acetaminophen) ≥ 15 days/month in the 3 months prior to Visit 1 per investigator's judgment
* Has a history of migraine aura with diplopia or impairment of level of consciousness, hemiplegic migraine, or retinal migraine as defined by ICHD-3
* A current diagnosis of chronic migraine as defined by ICHD-3 or a history of 15 or more headache days per month on average in the 6 months prior to Visit 1 in the investigator's judgment. A headache day is defined as a day in which there was any occurrence of a headache of a minimum duration of 2 hours or a headache of any duration for which acute medication was taken
* Has a current diagnosis of new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy as defined by ICHD-3
* Required hospital treatment of a migraine attack 3 or more times in the 6 months prior to Visit 1
* History of malignancy in the 5 years prior to Visit 1, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* History of any prior gastrointestinal conditions (eg, diarrhea syndromes, inflammatory bowel disease) that, per investigator judgment, may affect the absorption or metabolism of the study intervention; participants with prior gastric bariatric interventions (eg, Lap Band) which have been reversed are not excluded

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (73):
- United States (73):
  - Achieve Clinical Research, LLC /ID# 237098, Birmingham, Alabama
  - Barrow Neuro Institute /ID# 236775, Phoenix, Arizona
  - Arkansas Clinical Research /ID# 238032, Little Rock, Arkansas
  - California Headache and Balance Center /ID# 236247, Fresno, California
  - Sun Valley Research Center /ID# 236561, Imperial, California
  - Wr-Pri Llc /Id# 236007, Los Alamitos, California
  - Pharmacology Research Institute (PRI) - Newport Beach (Wake) /ID# 237691, Newport Beach, California
  - Excell Research, Inc /ID# 237721, Oceanside, California
  - George J. Rederich M.D. Inc. /ID# 235769, Torrance, California
  - Diablo Clinical Research /ID# 237570, Walnut Creek, California
  - Colorado Springs Neurological Associates (CSNA) /ID# 236556, Colorado Springs, Colorado
  - Advanced Neurosciences Research, LLC /ID# 237426, Fort Collins, Colorado
  - CNS Healthcare - Jacksonville /ID# 238245, Jacksonville, Florida
  - Health Awareness, Inc - Jupiter /ID# 236226, Jupiter, Florida
  - Suncoast Clinical Research /ID# 236934, New Port Richey, Florida
  - Sensible Healthcare /ID# 238090, Ocoee, Florida
  - Clinical Neuroscience Solutions, Inc /ID# 236608, Orlando, Florida
  - Accel Research Sites - St Petersburg Clinical Research Unit /ID# 237163, St. Petersburg, Florida
  - University of South Florida /ID# 234387, Tampa, Florida
  - ForCare Clinical Research /ID# 237092, Tampa, Florida
  - Premiere Research Institute - Palm Beach /ID# 238193, West Palm Beach, Florida
  - NeuroTrials Research Inc. /ID# 237365, Atlanta, Georgia
  - iResearch Atlanta, LLC /ID# 237390, Decatur, Georgia
  - Meridian Clinical Research (Neurology) - Savannah /ID# 234371, Savannah, Georgia
  - Clinical Research Atlanta - Headlands LLC /ID# 234438, Stockbridge, Georgia
  - Northwest Clinical Trials /ID# 234968, Boise, Idaho
  - Deaconess Clinic Downtown /ID# 236959, Evansville, Indiana
  - PMG Research of McFarland /ID# 238271, Ames, Iowa
  - Collective Medical Research /ID# 236402, Overland Park, Kansas
  - Kansas Institute of Research /ID# 236738, Overland Park, Kansas
  - Boston Clinical Trials /ID# 236559, Boston, Massachusetts
  - Michigan Headache & Neurological Institute (MHNI) /ID# 236565, Ann Arbor, Michigan
  - Minneapolis Clinic of Neurology - Golden Valley /ID# 238162, Golden Valley, Minnesota
  - Clinical Research Institute, Inc /ID# 238301, Minneapolis, Minnesota
  - StudyMetrix Research /ID# 236457, City of Saint Peters, Missouri
  - Clinvest Research LLC /ID# 237908, Springfield, Missouri
  - Princeton Center for Clinical Research /ID# 235734, Skillman, New Jersey
  - Bio Behavioral Health, Inc /ID# 238212, Toms River, New Jersey
  - Dent Neurosciences Research Center, Inc. /ID# 237039, Amherst, New York
  - Central New York Clinical Research /ID# 235694, Manlius, New York
  - Rochester Clinical Research /ID# 236842, New York, New York
  - Upstate Clinical Research Associates /ID# 238220, Williamsville, New York
  - PMG Research of Charlotte /ID# 237048, Charlotte, North Carolina
  - Raleigh Neurology Associates /ID# 237138, Raleigh, North Carolina
  - CTI Clinical Research Center /ID# 237278, Cincinnati, Ohio
  - University of Cincinnati /ID# 234403, Cincinnati, Ohio
  - Aventiv Research Columbus /ID# 236837, Columbus, Ohio
  - OK Clinical Research /ID# 236675, Edmond, Oklahoma
  - IPS Research Company /ID# 237674, Oklahoma City, Oklahoma
  - Summit Headlands LLC /ID# 236077, Portland, Oregon
  - Abington Neurological Associates - Abington /ID# 236257, Abington, Pennsylvania
  - Lehigh Center for Clinical Research /ID# 236703, Allentown, Pennsylvania
  - Suburban Research Associates - Media /ID# 236698, Media, Pennsylvania
  - Thomas Jefferson University Jefferson Headache Center /ID# 235821, Philadelphia, Pennsylvania
  - Frontier Clinical Research /ID# 237924, Smithfield, Pennsylvania
  - Clinical Trials of SC /ID# 237338, Charleston, South Carolina
  - WR-ClinSearch /ID# 238287, Chattanooga, Tennessee
  - CNS Healthcare - Memphis /ID# 236396, Memphis, Tennessee
  - FutureSearch Trials of Neurology /ID# 236428, Austin, Texas
  - Tekton Research, Inc. /ID# 237306, Austin, Texas
  - DiscoveResearch, Inc /ID# 236273, Bryan, Texas
  - FutureSearch Trials of Dallas, LP /ID# 236276, Dallas, Texas
  - Centex Studies, Inc. - Houston /ID# 237458, Houston, Texas
  - ClinPoint Trials /ID# 236618, Waxahachie, Texas
  - Advanced Research Institute /ID# 237749, Ogden, Utah
  - University of Utah /ID# 237602, Salt Lake City, Utah
  - Charlottesville Medical Research /ID# 237792, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc. (HRHR) /ID# 237253, Newport News, Virginia
  - Tidewater Integr Med Research /ID# 236867, Virginia Beach, Virginia
  - Sentara Neurology Specialists - Virginia Beach /ID# 234350, Virginia Beach, Virginia
  - Northwest Clinical Research Center /ID# 237585, Bellevue, Washington
  - Seattle Clinical Research Center /ID# 236912, Seattle, Washington
  - Puget Sound Neurology /ID# 236322, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Goadsby PJ, Jurgens TP, Brand-Schieber E, Nagy K, Liu Y, Boinpally R, Stodtmann S, Trugman JM. Efficacy of ubrogepant and atogepant in males and females with migraine: A secondary analysis of randomized clinical trials. Cephalalgia. 2025 Feb;45(2):3331024251320610. doi: 10.1177/03331024251320610. PMID 39982105
- [Derived] Schwedt TJ, Lipton RB, Goadsby PJ, Chiang CC, Klein BC, Hussar C, Liu C, Yu SY, Finnegan M, Trugman JM. Characterizing Prodrome (Premonitory Phase) in Migraine: Results From the PRODROME Trial Screening Period. Neurol Clin Pract. 2025 Feb;15(1):e200359. doi: 10.1212/CPJ.0000000000200359. Epub 2024 Oct 8. PMID 39399572
- [Derived] Lipton RB, Harriott AM, Ma JY, Smith JH, Stokes J, Gandhi P, Jariwala-Parikh K, Jensen GS, Trugman JM, Dodick DW. Effect of Ubrogepant on Patient-Reported Outcomes When Administered During the Migraine Prodrome: Results From the Randomized PRODROME Trial. Neurology. 2024 Sep 24;103(6):e209745. doi: 10.1212/WNL.0000000000209745. Epub 2024 Aug 28. PMID 39197113
- [Derived] Dodick DW, Goadsby PJ, Schwedt TJ, Lipton RB, Liu C, Lu K, Yu SY, Severt L, Finnegan M, Trugman JM. Ubrogepant for the treatment of migraine attacks during the prodrome: a phase 3, multicentre, randomised, double-blind, placebo-controlled, crossover trial in the USA. Lancet. 2023 Dec 16;402(10419):2307-2316. doi: 10.1016/S0140-6736(23)01683-5. Epub 2023 Nov 15. PMID 37979595
- See also: Additional information on study locations near you may be found at www.AllerganClinicalTrials.com. — https://www.allerganclinicaltrials.com/,http://www.investigatordatabank.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A: Participants randomized to Treatment Sequence A will receive placebo to treat their first qualifying prodrome event and ubrogepant 100 mg to treat their second qualifying prodrome event
  Ubrogepant 100mg: For each qualifying prodrome event, 2 compressed tablets containing 50 mg of ubrogepant will be taken orally when the participant is confident that a headache will follow within 1-6 hours
  Placebo: For each qualifying prodrome event, 2 compressed tablets containing placebo will be taken orally when the participant is confident that a headache will follow within 1-6 hours
- Treatment Sequence B: Participants randomized to Treatment Sequence B will receive ubrogepant 100 mg to treat their first qualifying prodrome event and placebo to treat their second qualifying prodrome event
  Ubrogepant 100mg: For each qualifying prodrome event, 2 compressed tablets containing 50 mg of ubrogepant will be taken orally when the participant is confident that a headache will follow within 1-6 hours
  Placebo: For each qualifying prodrome event, 2 compressed tablets containing placebo will be taken orally when the participant is confident that a headache will follow within 1-6 hours
Period: Overall Study
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started (Intent-to-Treat population consists of all randomized participants) | 264 | 254
Safety Population (Safety population consists of all treated participants who take at least 1 administration of study intervention) | 247 | 233
Completed | 223 | 215
Not Completed | 41 | 39
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 5 | 2
Not completed — Lack of Qualifying Event | 25 | 27
Not completed — Non-compliance with Study Drug | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population consists of all treated participants who take at least 1 administration of study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A | Treatment Sequence B | Total
Number analyzed (Participants) | 247 | 233 | 480
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (12.63) | 42.9 (13.10) | 42.3 (12.86)
Age, Customized [Count of Participants; unit: Participants]
  < 20 | 5 | 2 | 7
  20 - 29 | 42 | 38 | 80
  30 - 39 | 62 | 60 | 122
  40 - 49 | 68 | 64 | 132
  50 - 59 | 48 | 37 | 85
  60 - 69 | 18 | 28 | 46
  >= 70 | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 205 | 421
  Male | 31 | 28 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 32
  Not Hispanic or Latino | 229 | 216 | 445
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 22 | 15 | 37
  White | 214 | 209 | 423
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Absence of Headache of Moderate/Severe Intensity Within 24 Hours Post-dose
Description: The absence of a headache of moderate/severe intensity will be recorded by the participant in an electronic diary (eDiary) within 24 hours after taking double-blind study intervention during the prodrome in order to determine the attenuation of headache. The absence of moderate or severe headache are derived based on headache record and rescue use.
Time Frame: 24 hours after taking double-blind study intervention during the prodrome
Population: The Modified Intent-to-Treat (mITT) population consists of all randomized participants with at least 1 assessment of headache occurrence within 24 hours after taking double-blind study intervention for at least 1 qualifying prodrome event during the double-blind treatment period
Measure: Count of Participants; unit: Participants
Groups:
- Ubrogepant 100 mg: Ubrogepant 100mg: For each qualifying prodrome event, 2 compressed tablets containing 50 mg of ubrogepant will be taken orally when the participant is confident that a headache will follow within 1-6 hours
Arm/Group | Placebo | Ubrogepant 100 mg
Number analyzed (Participants) | 423 | 418
Participants | 121 | 190
Statistical Analysis 1: Comparison: Ubrogepant 100 mg; Test type: Superiority; p < .0001, generalized linear mixed model (GLMM); Odds Ratio (OR) = 2.09, 95% CI 2-sided [1.63 to 2.69]

2. Secondary Outcome: Percentage of Participants Reporting Absence of Headache of Moderate or Severe Intensity Within 48 Hours Post-dose
Description: The absence of a headache of moderate or severe intensity will be recorded by the participant in an eDiary within 48 hours after taking double-blind study intervention during the prodrome in order to determine the prevention of headache
Time Frame: 48 hours after taking double-blind study intervention during the prodrome
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ubrogepant 100 mg
Number analyzed (Participants) | 407 | 391
Participants | 100 | 159
Statistical Analysis 1: Comparison: Ubrogepant 100 mg; Test type: Superiority; p < .0001, generalized linear mixed model (GLMM); Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.63 to 2.78]

3. Secondary Outcome: Percentage of Participants Reporting Improvement in the Ability to Function Normally Over 24 Hours Post-dose
Description: The Functional Disability Scale (FDS) is a single item used to measure the participant's level to function normally. Participants will be asked to rate the performance of daily activities using 4 response options ranging from 0 (no disability, able to function normally) to 3 (severely impaired, cannot do all or most things, bed rest may be necessary) within 24 hours after taking double-blind study intervention during the prodrome
Time Frame: 24 hours after taking double-blind study intervention during the prodrome
Population: Modified Intent-to-Treat Population (randomized participants with at least 1 assessment of headache occurrence within 24 hours after taking double-blind study intervention for at least 1 qualifying prodrome event during the double-blind treatment period) with non-missing ability to function normally assessment at each timepoint after dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ubrogepant 100 mg
Number analyzed (Participants) | 449 | 448
Participants
  1 Hour: number analyzed (Participants) | 432 | 418
  1 Hour: Responder | 96 | 107
  1 Hour: Nonresponder | 336 | 311
  2 Hours: number analyzed (Participants) | 421 | 422
  2 Hours: Responder | 110 | 156
  2 Hours: Nonresponder | 311 | 266
  3 Hours: number analyzed (Participants) | 419 | 412
  3 Hours: Responder | 150 | 199
  3 Hours: Nonresponder | 269 | 213
  4 Hours: number analyzed (Participants) | 417 | 415
  4 Hours: Responder | 173 | 245
  4 Hours: Nonresponder | 244 | 170
  6 Hours: number analyzed (Participants) | 400 | 395
  6 Hours: Responder | 210 | 266
  6 Hours: Nonresponder | 190 | 129
  8 Hours: number analyzed (Participants) | 394 | 388
  8 Hours: Responder | 239 | 291
  8 Hours: Nonresponder | 155 | 97
  24 Hours: number analyzed (Participants) | 404 | 413
  24 Hours: Responder | 342 | 367
  24 Hours: Nonresponder | 62 | 46
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < .0001, generalized estimating equation (GEE); Geometric Mean Odds Ratio = 1.66, 95% CI 2-sided [1.40 to 1.96]

4. Secondary Outcome: Percentage of Participants Reporting Absence of Headache of Any Intensity Within 24 Hours Post-dose
Description: as for outcome 1
Time Frame: 24 hours after taking double-blind study intervention during the prodrome
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ubrogepant 100 mg
Number analyzed (Participants) | 439 | 434
Participants | 61 | 103
Statistical Analysis 1: Comparison: Ubrogepant 100 mg; Test type: Superiority; p < .0001, generalized linear mixed model (GLMM); Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.39 to 2.66]

ADVERSE EVENTS:
Time Frame: From first dose through 30 days after the last dose of study drug (approximately 30 days)
Description: Safety Population, all treated participants who take ≥1 administration of study intervention. Participants will be summarized according to the study intervention they actually received.
Arm/Group | Placebo | Ubrogepant 100 mg
All-Cause Mortality (participants affected / at risk) | 0/462 | 0/456
Serious Adverse Events (participants affected / at risk) | 1/462 | 0/456
Other Adverse Events (participants affected / at risk) | 35/462 | 50/456
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=462) | Ubrogepant 100 mg (N=456)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=462) | Ubrogepant 100 mg (N=456)
NAUSEA (Gastrointestinal disorders) | 17 (17) | 24 (25)
FATIGUE (General disorders) | 7 (7) | 12 (12)
DIZZINESS (Nervous system disorders) | 14 (14) | 11 (11)
SOMNOLENCE (Nervous system disorders) | 5 (5) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT04492020/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT04492020/SAP_001.pdf